CLINICAL TRIAL: NCT00935350
Title: Effect of Adding the Novel Fiber, PGX®,to Commonly Consumed Foods on Glycemic Response and Glycemic Index: A Practical and Effective Strategy for Reducing Post Prandial Blood Glucose Levels.
Brief Title: Reduction of the Glycemic Index by a Novel Viscous Polysaccharide
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Glycemic Index Laboratories, Inc (Industry)
Collaborators: InovoBiologic Inc. (Industry); Canadian Center for Functional Medicine (Other)
Responsible Party: Dr. Alexandra Jenkins, PhD, RD/ Vice President, Glycemic Index Laboratories, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GIL-6033
Record Dates: First submitted 2009-03-25; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Blood Glucose, Postprandial
Keywords: viscous; fibre; polysaccharide; blood glucose; postprandial
MeSH Terms: interventions — PolyGlycoplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (15):
- 1 (Placebo Comparator): Control White bread containing 50g available carbohydrate
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 2 (Placebo Comparator): White bread and milk control
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 3 (Placebo Comparator): Granola control
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 4 (Placebo Comparator): Cornflakes and milk control
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 5 (Placebo Comparator): White rice control
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 6 (Placebo Comparator): Fruit yogurt control
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 7 (Placebo Comparator): Turkey dinner control
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 8 (Experimental): Granola
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 9 (Experimental): Cornflakes and milk
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 10 (Experimental): White Rice
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 11 (Experimental): Fruit yogurt
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 12 (Experimental): Turkey dinner
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 13 (Placebo Comparator): White Bread
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 14 (Placebo Comparator): White bread
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- 15 (Experimental): Granola
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)

INTERVENTIONS:
Dietary Supplement: PolyGlycopleX (PGX) — 2.5 grams of PGX
  Arms: 15; 8
Dietary Supplement: PolyGlycopleX (PGX) — 5.0 grams of PGX
  Arms: 10; 11; 12; 8; 9
Dietary Supplement: PolyGlycopleX (PGX) — 0 grams of PGX
  Arms: 1; 13; 14; 2; 3; 4; 5; 6; 7

SUMMARY:
Reductions of postprandial glucose levels have been demonstrated previously with the addition of a novel viscous polysaccharide (NVP) to a glucose drink and standard white bread. This study explores whether these reductions are sustained when NVP is added to a range of commonly consumed foods.

DETAILED DESCRIPTION:
Recently, a commercial novel viscous polysaccharide (NVP)complex has been developed which is marketed in both the USA and Canada under the trade name PGX® (PolyGlycopleX) (InovoBiologic Inc, Calgary, AB, Canada). This complex consists of three viscous non starch polysaccharides which are processed using proprietary technology (EnviroSimplex®) to produce compressed granules which delays the onset of viscosity and increases palatability of the fiber when added to food. Previously, this fibre was shown to lower postprandial glucose levels in a dose responsive manner when mixed with a glucose drink and sprinkled onto a standard white bread demonstrating that the processing did not interfere with the effectiveness of the fiber. From this study the reduction in GI was calculated to be 7 units per gram of NVP when added to a solid food, however it is not known whether this relationship would be maintained when the NVP was added to a range of commonly eaten foods. This study therefore evaluates the effect of the addition or incorporation of NVP into a range of foods on postprandial glycemia and whether the reductions in glycemic index could be predicted using.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* 18-75 years old
* BMI less than 35 kg/m2

Exclusion Criteria:

* Medications influencing gastrointestinal function
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-05; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Relative Blood glucose response of food with and without NVP | Acute blood glucose response measured at 0, 15,30,45,60,90 and 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra L Jenkins, PhD, RD, Study Director — Glycemic Index Laboratories, Inc; Thomas MS Wolever, MD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jenkins AL, Kacinik V, Lyon M, Wolever TM. Effect of adding the novel fiber, PGX(R), to commonly consumed foods on glycemic response, glycemic index and GRIP: a simple and effective strategy for reducing post prandial blood glucose levels--a randomized, controlled trial. Nutr J. 2010 Nov 22;9:58. doi: 10.1186/1475-2891-9-58. PMID 21092221